CLINICAL TRIAL: NCT04773769
Title: Pilot Phase 2 Study of Graviola (Guanabana) Leaves for The Treatment of Patients With Relapsed or Refractory Gastric Adenocarcinoma, Adenocarcinoma of Gastroesophageal Junction, Hepatocellular Carcinoma, Pancreatic Adenocarcinoma, Low Grade Lymphomas and Colorectal Adenocarcinoma
Brief Title: Study of Guanábana Leaves for The Treatment of Patients With Gastric, Gastroesophageal Junction, Pancreatic and Colorectal Adenocarcinomas; Hepatocellular Carcinoma, and Low Grade Lymphomas
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Auxilio Mutuo Cancer Center (Other)
Responsible Party: Principal Investigator, Fernando Cabanillas, Medicine Doctor/Medical Director, Auxilio Mutuo Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCAM 18-01
Record Dates: First submitted 2018-12-04; First posted 2021-02-26 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Gastric Adenocarcinoma; Adenocarcinoma of the Gastroesophageal Junction; Hepatocellular Carcinoma; Pancreatic Adenocarcinoma; Low Grade Lymphoma; Colorectal Adenocarcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Overall Statistical design (Experimental): We will treat 9 patients of each tumor type with a tea made of Graviola Leaves. If no responses are observed then the trial will be closed for that particular histological type. Should a response occur, then the trial will continue to the second stage for that cell type until 24 patients are accrued. If 3 or more responses are observed out of 24 cases, then the result will be considered promising.
  Interventions: Dietary Supplement: Tea Made of Graviola Leaves

INTERVENTIONS:
Dietary Supplement: Tea Made of Graviola Leaves — Graviola leaves will be supplied to the patient with instructions on how to prepare the tea which will consist of 10 guanabana leaves which the patient will boil in 1 liter of water for 3 minutes. Once boiled, the formulation will be stores in the refrigerator and once cool enough the patient will start drinking 100 cc two times per day.
  The Treatment Period begins with Cycle 1 Day 1 dosing. Patients will take the tea continuously during a 28-day cycles, until there is an indication for treatment change based on response assessment.

SUMMARY:
Guanabana, known also as Graviola or Annona muricata is a tropical fruit which has been commonly used as complimentary/alternative medicine in Latin American countries. The main compounds in Graviola are the annonaceous acetogenins. These acetogenins have been shown to be selective and toxic against various types of cancer cells in-vitro and in-vivo experimental animal models. In spite of this evidence of anti tumor activity of Graviola, no prospective clinical studies have been carried out to determine if it also has clinical activity.The Investigator have observed two patients at Auxilio Mutuo Cancer Center who experienced significant tumor shrinkage while taking a tea made of Graviola leaves. Neither of these patients were taking any other treatment for their cancer. The investigator propose to conduct a study using guanabana leaves extract in patients with Gastroesophageal junction(GEJ) adenocarcinoma, as well as in Gastric adenocarcinoma, Hepatocellular carcinoma, Pancreatic adenocarcinoma, Low Grade Lymphomas and Colorectal adenocarcinoma.

DETAILED DESCRIPTION:
Patients with relapsed/refractory gastric adenocarcinoma, adenocarcinoma of gastroesophageal junction, hepatocellular carcinoma, colorectal adenocarcinoma will be eligible. Colorectal adenocarcinomas will be eligible after failing second line therapy while the remainder will be eligible after first line therapy depending on the judgment of the treating oncologist. Any patient who refuse to receive chemotherapy will also be eligible even if they have not received chemotherapy. Patients with low grade lymphomas including chronic lymphocytic leukemias whose favorable blood counts and lack of symptoms make the candidates for "watch and wait" approach as well as any patient with low grade lymphoma who because of age or co-morbidity might not be eligible for chemotherapy or who refuse chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign an informed consent form.
* Age > 18 years at the time of signing the informed consent form.
* Willing and able to adhere to the study visit schedule and other protocol requirements.
* Must have measurable or evaluable disease.
* All previous cancer therapy, including radiation, hormonal therapy and surgery, must have been discontinued at least 2 weeks prior to treatment in this study.
* Performance status of ≤ 2 on the Eastern Cooperative Oncology Group (ECOG) scale at study entry.

Exclusion Criteria:

* Patients actively taking guanabana or guanabana tea daily or who have used it at some point after their diagnosis of cancer.
* Patients with Parkinson's disease.
* Serum Total Bilirubin ≥ 3.0 mg/dL
* Serum Creatinine level ≥ 3.0 mg/dL
* Central Nervous System (CNS) involvement.
* Known human immunodeficiency virus (HIV) infection; Known active hepatitis B or hepatitis C infection.
* Females who are pregnant (positive urine test) or breast-feeding females.
* Any history of a medical condition or a concomitant medical condition that, in the opinion of the investigator, would compromise the subject's ability to safely complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2018-11-07 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
RECIST criteria | Through study completion, an average of 3 years.
  RECIST criteria will be used to measure response in solid tumors.
Cheson criteria | Through study completion, an average of 3 years.
  Cheson criteria will be used for lymphomas.
Blood Counts | Through study completion, an average of 3 years.
  Cases with Chronic Lymphocytic Leukemia will have their Complete Blood Counts monitored and the Absolute lymphocyte count will be followed for response.

CONTACTS AND LOCATIONS:
Overall Officials: Fernado Cabanillas, MD, Principal Investigator — Hospital Español Auxilio Mutuo Inc.
Locations (1):
- Auxilio Mutuo Cancer Center, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chamcheu JC, Rady I, Chamcheu RN, Siddique AB, Bloch MB, Banang Mbeumi S, Babatunde AS, Uddin MB, Noubissi FK, Jurutka PW, Liu YY, Spiegelman VS, Whitfield GK, El Sayed KA. Graviola (Annona muricata) Exerts Anti-Proliferative, Anti-Clonogenic and Pro-Apoptotic Effects in Human Non-Melanoma Skin Cancer UW-BCC1 and A431 Cells In Vitro: Involvement of Hedgehog Signaling. Int J Mol Sci. 2018 Jun 16;19(6):1791. doi: 10.3390/ijms19061791. PMID 29914183
- [Background] Deep G, Kumar R, Jain AK, Dhar D, Panigrahi GK, Hussain A, Agarwal C, El-Elimat T, Sica VP, Oberlies NH, Agarwal R. Graviola inhibits hypoxia-induced NADPH oxidase activity in prostate cancer cells reducing their proliferation and clonogenicity. Sci Rep. 2016 Mar 16;6:23135. doi: 10.1038/srep23135. PMID 26979487
- [Background] Magadi VP, Ravi V, Arpitha A, Litha, Kumaraswamy K, Manjunath K. Evaluation of cytotoxicity of aqueous extract of Graviola leaves on squamous cell carcinoma cell-25 cell lines by 3-(4,5-dimethylthiazol-2-Yl) -2,5-diphenyltetrazolium bromide assay and determination of percentage of cell inhibition at G2M phase of cell cycle by flow cytometry: An in vitro study. Contemp Clin Dent. 2015 Oct-Dec;6(4):529-33. doi: 10.4103/0976-237X.169863. PMID 26681860
- [Background] Paul J, Gnanam R, Jayadeepa RM, Arul L. Anti cancer activity on Graviola, an exciting medicinal plant extract vs various cancer cell lines and a detailed computational study on its potent anti-cancerous leads. Curr Top Med Chem. 2013;13(14):1666-73. doi: 10.2174/15680266113139990117. PMID 23889049
- [Background] Sun S, Liu J, Kadouh H, Sun X, Zhou K. Three new anti-proliferative Annonaceous acetogenins with mono-tetrahydrofuran ring from graviola fruit (Annona muricata). Bioorg Med Chem Lett. 2014 Jun 15;24(12):2773-6. doi: 10.1016/j.bmcl.2014.03.099. Epub 2014 Apr 18. PMID 24780120
- [Background] Sun S, Liu J, Zhou N, Zhu W, Dou QP, Zhou K. Isolation of three new annonaceous acetogenins from Graviola fruit (Annona muricata) and their anti-proliferation on human prostate cancer cell PC-3. Bioorg Med Chem Lett. 2016 Sep 1;26(17):4382-5. doi: 10.1016/j.bmcl.2015.06.038. Epub 2015 Jun 25. PMID 27499453
- [Background] Yang C, Gundala SR, Mukkavilli R, Vangala S, Reid MD, Aneja R. Synergistic interactions among flavonoids and acetogenins in Graviola (Annona muricata) leaves confer protection against prostate cancer. Carcinogenesis. 2015 Jun;36(6):656-65. doi: 10.1093/carcin/bgv046. Epub 2015 Apr 11. PMID 25863125
- [Background] Torres MP, Rachagani S, Purohit V, Pandey P, Joshi S, Moore ED, Johansson SL, Singh PK, Ganti AK, Batra SK. Graviola: a novel promising natural-derived drug that inhibits tumorigenicity and metastasis of pancreatic cancer cells in vitro and in vivo through altering cell metabolism. Cancer Lett. 2012 Oct 1;323(1):29-40. doi: 10.1016/j.canlet.2012.03.031. Epub 2012 Apr 1. PMID 22475682
- [Background] Li Y, Ye J, Chen Z, Wen J, Li F, Su P, Lin Y, Hu B, Wu D, Ning L, Xue Q, Gu H, Ning Y. Annonaceous acetogenins mediated up-regulation of Notch2 exerts growth inhibition in human gastric cancer cells in vitro. Oncotarget. 2017 Mar 28;8(13):21140-21152. doi: 10.18632/oncotarget.15502. PMID 28416750
- [Background] Prabhakaran K, Ramasamy G, Doraisamy U, Mannu J, K R, Murugesan JR. Polyketide Natural Products, Acetogenins from Graviola (Annona muricata L), its Biochemical, Cytotoxic Activity and Various Analyses Through Computational and Bio-Programming Methods. Curr Pharm Des. 2016;22(34):5204-5210. doi: 10.2174/1381612822666160531163144. PMID 27262333
- [Background] Caparros-Lefebvre D, Elbaz A. Possible relation of atypical parkinsonism in the French West Indies with consumption of tropical plants: a case-control study. Caribbean Parkinsonism Study Group. Lancet. 1999 Jul 24;354(9175):281-6. doi: 10.1016/s0140-6736(98)10166-6. PMID 10440304
- [Background] Hollerhage M, Rosler TW, Berjas M, Luo R, Tran K, Richards KM, Sabaa-Srur AU, Maia JG, Moraes MR, Godoy HT, Hoglinger GU, Smith RE. Neurotoxicity of Dietary Supplements from Annonaceae Species. Int J Toxicol. 2015 Nov-Dec;34(6):543-50. doi: 10.1177/1091581815602252. Epub 2015 Sep 24. PMID 26405269
- [Background] Simon R. Optimal two-stage designs for phase II clinical trials. Control Clin Trials. 1989 Mar;10(1):1-10. doi: 10.1016/0197-2456(89)90015-9. PMID 2702835
- [Background] Lannuzel A, Hoglinger GU, Champy P, Michel PP, Hirsch EC, Ruberg M. Is atypical parkinsonism in the Caribbean caused by the consumption of Annonacae? J Neural Transm Suppl. 2006;(70):153-7. doi: 10.1007/978-3-211-45295-0_24. PMID 17017523
- [Background] Therasse P, Arbuck SG, Eisenhauer EA, Wanders J, Kaplan RS, Rubinstein L, Verweij J, Van Glabbeke M, van Oosterom AT, Christian MC, Gwyther SG. New guidelines to evaluate the response to treatment in solid tumors. European Organization for Research and Treatment of Cancer, National Cancer Institute of the United States, National Cancer Institute of Canada. J Natl Cancer Inst. 2000 Feb 2;92(3):205-16. doi: 10.1093/jnci/92.3.205. PMID 10655437
- See also: Graviola: A Systematic Review on Its Anticancer Properties — https://www.researchgate.net/profile/Ioannis_Patrikios/publication/290448944_Graviola_A_Systematic_Review_on_Its_Anticancer_Properties/Links/5699700308ae6169e5518da2.pdf